CLINICAL TRIAL: NCT07206602
Title: A Pilot Study Assessing Outcomes Of Artificial Intelligence-Guided Left Bundle Branch Area Pacing For Cardiac Resynchronization In Heart Failure
Brief Title: AI-Guided Left Bundle Branch Area Pacing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Fatima M. Ezzeddine, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 25-007700
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- AI-guided (Experimental)
  Interventions: Device: AI-assisted Left Bundle Branch Area Pacing
- Control (Active Comparator)
  Interventions: Procedure: Left Bundle Branch Area Pacing

INTERVENTIONS:
Device: AI-assisted Left Bundle Branch Area Pacing — Patients will undergo a Left Bundle Branch Area Pacing (LBBAP) procedure using AI assisted technology
  Arms: AI-guided
Procedure: Left Bundle Branch Area Pacing — Patients will undergo a Left Bundle Branch Area Pacing (LBBAP) procedure
  Arms: Control

SUMMARY:
The purpose of this study is to compare the effectiveness of AI-guided LBBAP versus conventional LBBAP (not AI-guided) in improving CRT response rates and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria

* Age: 18 years or older.
* Left Ventricular Ejection Fraction (LVEF): <50% within 6 months prior to enrollment.
* QRS Duration: Resting QRS duration ≥ 130 ms on ECG OR anticipated right ventricular pacing > 40% OR device in place with right ventricular pacing > 40% within 6 months prior to enrollment.
* Medical Therapy: Optimized on guideline-directed medical therapy for heart failure.
* AI-ECG probability of low LVEF: >0.5

Exclusion Criteria

* Age less than 18 years old
* Inability to follow-up
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
CRT response rate | Baseline, 6 months
  CRT response is defined as an absolute increase of >5% in left ventricular ejection fraction (LVEF) after 6 months of CRT

SECONDARY OUTCOMES:
NYHA (New York Heart Association) Class | Baseline, 6 months
  The New York Heart Association (NYHA) classification will be assessed using the NYHA questionnaire, which evaluates the extent of physical limitations caused by heart failure. This system categorizes patients into one of four classes, with higher classes indicating more severe functional impairment.
Number of Hospitalizations | 6 months
  Number of Hospitalizations will be determined by the number of participants that are hospitalized for heart failure.
Number of Deaths | 6 months
  Number of patient deaths by any cause
Left Ventricular Linear Dimensions | Baseline, 3 months
  Left Ventricular Linear Dimensions will be measured by an echocardiogram. A lower value indicates better cardiac function.
Left Ventricular Linear Volume | Baseline, 3 months
  Left Ventricular Linear Volume will be measured by an echocardiogram. A lower value indicates better cardiac function.
Procedural success: LBBAP-conventional arm | Baseline
  LBBAP is considered successful if unipolar paced QRS morphology demonstrated a Qr or qR morphology in lead V1 along with any 1 of the following criteria:
  * Left bundle branch potential
  * Transition to selective left bundle branch capture or left ventricular septal capture during threshold testing or programmed stimulation
  * R-wave peak time <90 ms in V5-V6
  * V6-V1 interpeak interval >44 ms
Procedural success: AI-LBBAP arm | Baseline
  Procedural success is defined as improvement in the AI-ECG predicted likelihood of having a low LVEF from greater than 0.5 at baseline to less than 0.5 after LBBAP.
Fluoroscopy time | Baseline, Approximately 30 minutes
  Fluoroscopy time will be determined by the amount of time that fluoroscopy is used to guide the left bundle branch area pacing (an average of 30 minutes)
Total procedure time | Baseline, Approximately 1-2 hours
  Total procedure time will be determined by the start of the LBBAP procedure until completion (an average of 2 hours)
Lead pacing thresholds | Baseline
  Lead pacing thresholds will be measured in Voltage at millisecond.
Impedance | Baseline
  Impedance will be measured in Ohms.
Sensing Parameters | Baseline
  Sensing Parameters will be measured in mV (milliVolts)

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Ezzeddine, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No